CLINICAL TRIAL: NCT02160834
Title: A Mobile Health Approach to Reducing Sedentary Time in Bariatric Surgery Patients
Brief Title: Reducing Sedentary Time in Obese Adults (Study 2)
Acronym: B-MOBILE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not initiated
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03KD095740-02; R03DK095740 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
Keywords: Sedentary behavior; Physical activity; Obesity; Mobile health; Smartphone; Time spent sedentary
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B-MOBILE smartphone-based intervention (3-min break) (Experimental): Participants will receive a smartphone with B-MOBILE app that automatically monitors their sedentary time and prompts them after every 30 continuous sedentary minutes to walk for at least 3 minutes. Participants who meet this goal will receive reinforcing feedback in "real time."
  Interventions: Behavioral: B-MOBILE Smartphone-Based Intervention (3-min break)
- B-MOBILE Smartphone-Based Intervention (6-min break) (Experimental): Participants will receive a smartphone with B-MOBILE app that automatically monitors their sedentary time and prompts them after every 60 continuous sedentary minutes to walk for at least 6 minutes. Participants who meet this goal will receive reinforcing feedback in "real time."
  Interventions: Behavioral: B-MOBILE Smartphone-Based Intervention (6-min break)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: B-MOBILE Smartphone-Based Intervention (3-min break) — Participants will receive a smartphone with B-MOBILE app that automatically monitors their sedentary time and prompts them after every 30 continuous sedentary minutes to walk for at least 3 minutes. Participants who meet this goal will receive reinforcing feedback in "real time."
  Arms: B-MOBILE smartphone-based intervention (3-min break)
Behavioral: B-MOBILE Smartphone-Based Intervention (6-min break) — Participants will receive a smartphone with B-MOBILE app that automatically monitors their sedentary time and prompts them after every 60 continuous sedentary minutes to walk for at least 6 minutes. Participants who meet this goal will receive reinforcing feedback in "real time."
  Arms: B-MOBILE Smartphone-Based Intervention (6-min break)

SUMMARY:
Greater time spent in sedentary behaviors, independent of physical activity level, can increase risk of morbidity and mortality. Objective assessments indicate that bariatric surgery patients spend large amounts of time in sedentary behaviors. The present study is the first to test whether a mobile health (mHealth) approach that employs widely adopted smartphone technology to monitor and modify sedentary behaviors as they occur is a feasible and acceptable method of reducing sedentary time in these patients and other obese populations.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery patients and other obese individuals will be considered
* Body mass index >= 25 kg/m2

Exclusion Criteria:

* Report being unable to engage in daily activities and walk continuously for >= 10 minutes without assistance
* Are currently involved in a physical activity intervention.
* Are unable to read or understand the study materials
* Are currently taking medications that cause dizziness and/or feeling faint when sitting or standing.
* Report any condition that in the opinion of investigators would preclude adherence to the intervention protocol including plans to relocate, history of substance abuse or other significant psychiatric problems, or terminal illness.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in percentage of daily sedentary time from baseline to post-intervention. | 8 weeks

SECONDARY OUTCOMES:
Change in percentage of daily sedentary time from baseline to follow-up | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dale S Bond, PhD, Principal Investigator — The Miriam Hospital/Brown Alpert Medical School
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States